CLINICAL TRIAL: NCT06779201
Title: Study on the Effect and Mechanism of Fasting on Human Metabolism and Immunity
Brief Title: Fasting Effects on Metabolism and Immunity Study in Human
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: fasting
Record Dates: First submitted 2025-01-05; First posted 2025-01-16 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Fasting
Keywords: Fasting; Metabolism; Immunity; Brain function; Intestinal flora
MeSH Terms: conditions — Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adults who can tolerate a certain degree of hunger (Experimental): The subjects will undergo a complete fast for one week (water is allowed).
  Interventions: Other: Fasting

INTERVENTIONS:
Other: Fasting — One-week fasting without limit of water drink (Participants can feel free to drink water )

SUMMARY:
This study aims to investigate the effects of 1-week fasting but not prohibiting water drink on human immune function, metabolic indicators, and brain function in human, and to explore the underlying mechanisms of these changes from a multi-omics perspective and/or other ways.

DETAILED DESCRIPTION:
As a historic practice, fasting has a place in religion, culture and modern medicine. In recent years, studies have found that moderate food interruption can positively affect metabolism, immunity, and brain function. It can promote cellular autophagy, improve insulin sensitivity, reduce inflammation, and may protect brain health. Intermittent fasting is thought to improve metabolic health, reduce the risk of obesity and type 2 diabetes, and promote cellular self-repair by regulating signaling pathways. Food fasting also improves insulin sensitivity, reduces blood glucose, reduces inflammatory markers, and improves fat oxidation rate, contributing in the prevention and treatment of metabolic diseases. Moreover, food fasting can regulate immune cell function, reduce chronic inflammation, and may regulate immune function by affecting gut microbiota diversity. In terms of brain function, fasting may improve cognitive function by promoting neuroplasticity and enhancing neuroprotective mechanisms. However, most of the existing studies focus on animal experiments, lack large-scale human clinical trials, and the mechanism of feeding is not completely clear. This study will explore the effects of complete fasting for 1 week (but can feel free to drink water) on human immune function, metabolic indicators and brain function in human, and analyze its change mechanism from a multi-omics perspective and/or other ways, so as to provide new data support for understanding the biological mechanism of fasting, and promote its application in disease prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old, gender is not limited;
2. BMI≥18.5;
3. Can tolerate a certain degree of hunger;
4. Can voluntarily sign written informed consent.

Exclusion Criteria:

1. Women planning pregnancy, pregnancy and breastfeeding;
2. Previous liver disease, chronic kidney disease, heart disease and cerebrovascular disease;
3. Suffering from acute infectious diseases or chronic wasting diseases;
4. Have used antibiotic drugs in the past 3 months, and have used prebiotic or probiotic supplements or products in the past month;
5. Participate in other clinical investigators within 3 months before enrollment in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of cytokine levels in subjects' blood (and/or urine/stool) samples from T1 to T2, T3, T4, and T5. | T1 (Baseline/Pre-fasting): Day 0; T2 (End of one week fasting): Day 8; T3 (End of one week re-feeding): Day 15; T4 (End of four weeks re-feeding): Day 36; T5 (End of twelve weeks re-feeding): Day 92.
  Cytokines measured included pro-inflammatory cytokines such as IL-1β, IL-6, and TNF-α, as well as anti-inflammatory cytokines such as IL-10 and TGF-β.
The change of metabolite levels in subjects' blood (and/or urine/stool) samples from T1 to T2, T3, T4, and T5. | T1 (Baseline/Pre-fasting): Day 0; T2 (End of one week fasting): Day 8; T3 (End of one week re-feeding): Day 15; T4 (End of four weeks re-feeding): Day 36; T5 (End of twelve weeks re-feeding): Day 92.
  Metabolites measured include metabolic levels of amino acids, short-chain fatty acids, steroid hormones, fat-soluble vitamins, and other substances.

SECONDARY OUTCOMES:
The change in concentration of intestinal flora species，rate of change in bacterial diversity，abundance of functional genes in subjects' stool samples from T1 to T2, T3, T4, and T5. | T1 (Baseline/Pre-fasting): Day 0; T2 (End of one week fasting): Day 8; T3 (End of one week re-feeding): Day 15; T4 (End of four weeks re-feeding): Day 36; T5 (End of twelve weeks re-feeding): Day 92.
  Measure the concentration of specific bacterial species, e.g., relative and absolute abundance of Thick-walled phylum, Mycobacterium phylum, etc.; assess the rate of change in the diversity of the bacterial community, including α-diversity and β-diversity.
The change of brain function from T1 to T2, T3, T4, and T5. | T1 (Baseline/Pre-fasting): Day 0; T2 (End of one week fasting): Day 8; T3 (End of one week re-feeding): Day 15; T4 (End of four weeks re-feeding): Day 36; T5 (End of twelve weeks re-feeding): Day 92.
  The effects of fasting on brain function were assessed by resting-state functional magnetic resonance imaging (rs-fMRI) and diffusion tensor imaging (DTI) for local coherence (ReHo) and low-frequency amplitude (ALFF), which were used to assess changes in functional brain activity. Fraction of anisotropy (FA), axial dispersion (AD), radial dispersion (RD), and mean dispersion (MD), were used to assess the structural integrity of cerebral white matter.
The change of blood lipid levels from T1 to T2, T3, T4, and T5. | T1 (Baseline/Pre-fasting): Day 0; T2 (End of one week fasting): Day 8; T3 (End of one week re-feeding): Day 15; T4 (End of four weeks re-feeding): Day 36; T5 (End of twelve weeks re-feeding): Day 92.
  Lipids measured include total cholesterol, triglycerides, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, Apolipoprotein A, and Apolipoprotein B.
The change of homocysteine levels from T1 to T2, T3, T4, and T5 | T1 (Baseline/Pre-fasting): Day 0; T2 (End of one week fasting): Day 8; T3 (End of one week re-feeding): Day 15; T4 (End of four weeks re-feeding): Day 36; T5 (End of twelve weeks re-feeding): Day 92.
The change of insulin levels in subjects' blood samples from T1 to T2, T3, T4, and T5. | T1 (Baseline/Pre-fasting): Day 0; T2 (End of one week fasting): Day 8; T3 (End of one week re-feeding): Day 15; T4 (End of four weeks re-feeding): Day 36; T5 (End of twelve weeks re-feeding): Day 92.
The change of thyroid function level from T1 to T2, T3, T4, and T5. | T1 (Baseline/Pre-fasting): Day 0; T2 (End of one week fasting): Day 8; T3 (End of one week re-feeding): Day 15; T4 (End of four weeks re-feeding): Day 36; T5 (End of twelve weeks re-feeding): Day 92.
  Thyroid function indicators measured include thyroid-stimulating hormone (TSH), free triiodothyronine (FT3), free thyroxine (FT4), total triiodothyronine (TT3), total thyroxine (TT4), antithyroid peroxidase antibody (TPOAb), antithyroglobulin antibody (TGAb), and thyrotropin receptor antibody (TRAb).
The change of body fat percentage from T1 to T2, T3, T4, and T5. | T1 (Baseline/Pre-fasting): Day 0; T2 (End of one week fasting): Day 8; T3 (End of one week re-feeding): Day 15; T4 (End of four weeks re-feeding): Day 36; T5 (End of twelve weeks re-feeding): Day 92.

CONTACTS AND LOCATIONS:
Overall Officials: Hongxing Wang, MD & PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No